CLINICAL TRIAL: NCT06867523
Title: The Effect of Eye Masks and Earplugs on Delirium and Pain Prevention in Pediatric Intensive Care Unit Patients
Brief Title: Eye Masks and Earplugs for Delirium and Pain Prevention in Pediatric Intensive Care Unit
Acronym: PICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Şenay ARAS DOĞAN, Asst. Prof. Dr., Bozok University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023-14/15; THD-2025-1489 (Other Grant/Funding Number: Bozok University Scientific Research Projects Unit (BAP))
Record Dates: First submitted 2025-03-05; First posted 2025-03-10 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Pain Management; Pediatric Intensive Care Unit; Non-Pharmacological Interventions; Critical Care Nursing; Pediatric Delirium
Keywords: Pediatric Intensive Care; Non-Pharmacological Interventions; Delirium Prevention; Pain Management; Critical Care Nursing
MeSH Terms: conditions — Agnosia | interventions — Ear Protective Devices

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to an intervention group (eye mask and earplugs) or a control group (standard nursing care).
Who Masked: Participant, Care Provider
Masking Description: This study follows a double-blind design. Participants (patients) and care providers (nurses) are blinded to group assignments. However, outcome assessors (who are also nurses) may become aware of group allocations while assessing delirium and pain scores. The principal investigator is aware of the group assignments to ensure protocol adherence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eye Mask & Earplugs (Experimental): Participants in this group will use an eye mask and earplugs between 11:00 PM and 07:00 AM for three consecutive nights. The goal is to reduce environmental stimuli and evaluate the effects on delirium incidence and pain levels.
  Interventions: Other: Eye Mask; Other: Earplugs
- Standard Nursing Care (No Intervention): Participants in this group will receive standard nursing care without the use of an eye mask or earplugs. Their delirium incidence and pain levels will be assessed under usual care conditions.

INTERVENTIONS:
Other: Eye Mask — Participants in this group will wear an eye mask between 11:00 PM and 07:00 AM for three consecutive nights to assess its effects on delirium and pain levels in pediatric intensive care unit patients
  Arms: Eye Mask & Earplugs
Other: Earplugs — Participants in this group will use earplugs between 11:00 PM and 07:00 AM for three consecutive nights to evaluate their effects on delirium incidence and pain levels.
  Arms: Eye Mask & Earplugs

SUMMARY:
This randomized controlled clinical trial aims to evaluate the effect of nighttime application of eye masks and earplugs on the incidence of delirium and pain levels in pediatric intensive care unit (PICU) patients aged 6-12 years.

Research Questions

This study seeks to answer the following key questions:

Do eye masks and earplugs reduce the incidence of delirium compared to standard nursing care in PICU patients? Do eye masks and earplugs lower pain levels compared to standard nursing care in PICU patients? Study Design

Participants will be randomly assigned to one of the following groups:

Intervention Group: Participants will wear an eye mask and earplugs from 11:00 PM to 07:00 AM for three consecutive nights.

Control Group: Participants will receive standard nursing care without any interventions.

Both groups will be assessed daily at 08:00 AM using the following standardized measures:

Cornell Pediatric Delirium Scale (to assess symptoms of confusion and disorientation) Validated faces-based pediatric pain scale via a secure telehealth platform (to measure pain levels) Glasgow Coma Scale (GCS) (to evaluate consciousness levels) Significance and Impact This study investigates the impact of reducing environmental stimuli (light and noise) on delirium incidence and pain levels in critically ill pediatric patients. The findings may contribute to the development of non-pharmacological interventions aimed at improving patient comfort and care in intensive care settings.

Data Analysis Statistical analyses will be performed using SPSS (version 27) to compare delirium incidence and pain levels between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 6 and 12 years.
* Receiving treatment in the Pediatric Intensive Care Unit (PICU).
* Expected to stay in the intensive care unit for more than 24 hours.
* Having a Glasgow Coma Scale (GCS) score of 9 or above.
* Not receiving sedation.

Exclusion Criteria:

* Children with diagnosed intellectual, auditory, or visual impairments.
* Children with a psychiatric diagnosis.
* Patients using hearing aids.
* Patients diagnosed with brain tumors.
* Patients requiring mechanical ventilation.
* Patients using benzodiazepines or other strong sedative medications.
* Patients with an expected ICU stay of fewer than three days.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2024-08-25 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Delirium in Pediatric ICU Patients | 3 days after intervention
  Delirium incidence will be assessed using the Cornell Pediatric Delirium Scale every morning at 08:00 AM for three consecutive days. The nurse rates each item of the screening questions on a scale from 0 (lowest) to 4 (highest). Scores ≥9 indicate delirium.
Pain Levels in Pediatric ICU Patients | 3 days after intervention
  Pain levels will be assessed every morning at 08:00 AM for three consecutive days using a validated faces-based pediatric pain assessment tool administered via a secure telehealth platform.

CONTACTS AND LOCATIONS:
Locations (1):
- Bozok University, Yozgat, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided